CLINICAL TRIAL: NCT00198042
Title: Bone Tunnel Widening Following ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Inion Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22129
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Anterior Cruciate Ligament Injury; Knee Injuries
Keywords: ACL; Tunnel; Widening
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

ARMS (1):
- Surgical Reconstruction of the ACL (Experimental)
  Interventions: Procedure: Surgical reconstruction of the ACL

INTERVENTIONS:
Procedure: Surgical reconstruction of the ACL — Surgical reconstruction of the ACL

SUMMARY:
Hypothesis 1: There is less tunnel-widening with bone-patella tendon-bone graft compared with the hamstring graft when the same fixation method is used. Tunnel widening is greater with achilles tendon allografts versus autograft bone-patella tendon-bone and hamstring autografts.

Hypothesis 2: Tunnel widening occurs in the early post-operative period (< 8 weeks) when the tendon remodels within the bone tunnels.

Hypothesis 3: Low pre-operative bone mineral density is associated with tunnel widening.

DETAILED DESCRIPTION:
This will be a prospective study for patients undergoing ACL reconstruction using bone-patella tendon-bone graft, hamstring graft or achilles allograft. Each group will have ACL reconstruction with fixation using bioabsorbable interference screws on the femoral and tibial side. Patients will be evaluated on the day of surgery, 6, 12, 24, 52 and 104 weeks post-operatively. Evaluations will include pre-operative regional and standard bone mineral density measurements, post-operative MRI evaluation of tunnel dimensions and bone-tendon interface, radiographic evaluation of tunnel dimensions and routine clinical follow-up.

Interventions or Observations - outline specific procedures, treatments and/or interventions, as well as sources of research material to be utilized, which will involve human subjects or human materials that will be part of this research project.

This study will require a pre-operative bone mineral density measurement in the Nuclear Medicine Division of the Department of Radiology at HSS. Standard measurements of the femoral neck, spine as well as regional studies of the distal femur and proximal tibia of the injured knee will be performed.

On the day of surgery, the patient will undergo ACL reconstruction using bioabsorbable interference screw fixation of the hamstring, bone-patella tendon-bone graft, or achilles allograft. This is a standard procedure. The choice of graft type (hamstring, bone-patella tendon-bone graft, or achilles allograft) will be discussed with the patients and the patient will decide graft type pre-operatively. In this study, we will standardize the fixation method by using bioabsorbable interference screws. Post-operatively, the patient will undergo a limited MRI scan to evaluate the tunnel dimensions as well as graft placement prior to discharge from the hospital.

During the patients' 6 weeks, 12 weeks and 24 weeks clinical follow-up, they will be evaluated by their orthopaedic surgeon for clinical progress. Standard radiographs will be obtained of the patient's knee at the 6 weeks and 24 weeks follow-up visit. These are standard radiographic evaluations and are of no additional charge to the patients. We will utilize these images for radiographic measurements of tunnel expansion. During these visits, the patients will also undergo limited MRI scan of the femoral tunnel and tibia tunnel. With the serial MRI images, we will be able to make accurate measurements of the femoral and tibial tunnels. In addition, we will be able to evaluate the bone-tendon interface as well as the maturation of the intra-articular portion of the ACL graft. At 24, 52 and 104 weeks the patients will also be given standard IKDC and Lysholm clinical knee outcome questionnaires and will have objective stability measurements of both the operative and non-operative knees using a KT-1000 instrument.

Overall Study Protocol:

Pre-operative work-up

1. Bone mineral density measurement by D.E.X.A.

Day of Surgery:

1. ACL reconstruction using bioabsorbable interference screws
2. Limited CT scans to quantitate tunnel dimensions

6 weeks post-operatively

1. Regular clinical follow-up
2. Regular plain radiographs to quantitate tunnel dimensions
3. Limited MRI scans to quantitate tunnel dimensions

12 weeks post-operatively

1. Regular clinical follow-up
2. Limited MRI scans to quantitate tunnel dimensions

24 weeks post-operatively

1. Regular clinical follow-up and KT-1000 measurements
2. Regular plain radiographs to quantitate tunnel dimensions
3. MRI study to evaluate tendon-bone interface, graft maturation, tunnel dimensions and trabecular remodeling
4. Patients will answer IKDC and Lysholm knee questionnaires

52 weeks post-operatively

1. Regular clinical follow-up and KT-1000 measurements
2. Patients will answer IKDC and Lysholm knee questionnaires
3. Limited MRI

104 weeks post-operatively

1. Regular clinical follow-up and KT-1000 measurements
2. Patients will answer IKDC and Lysholm knee questionnaires
3. Limited MRI

Number of Subjects (power justification for numbers)

A power analysis was performed to determine the number of subjects needed to determine significance between the hamstring and bone-patella tendon-bone group. Data from previous studies demonstrate tunnel widening up to 77 ± 28% following ACL reconstruction using hamstring tendons. We estimate that a 30% decrease in this amount of tunnel widening would be clinically significant. This extrapolates to a 54% increase in tunnel dimensions. Using these estimations, a power of 0.80 with α = 0.5 is achieved using 20 subjects per group (BPTB versus hamstring).

ELIGIBILITY:
Inclusion Criteria:

* Individuals within the age range of 18 to 55 years who are diagnosed with anterior cruciate insufficiency and have decided to undergo ACL reconstruction using autogenous graft will be included in the study.

Exclusion Criteria:

* Individuals that have previous knee surgeries, multi-ligament injuries, systemic ligament disorders such as Ehlers Danlos syndrome or connective tissue disorders will be excluded from the study.
* Individuals who are pregnant or expect to be pregnant during the course of the study or who are especially concerned with X-ray exposure should also be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2004-06; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rodeo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from one surgeons practice.
Groups:
- Patients: Eighteen patients (including 12 men), mean age 35.5 6 8.7 years, who underwent ACL reconstruction.
Period: Overall Study
Arm/Group | Patients
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants] — Age, categorical
  Participants
    <=18 years | 0
    Between 18 and 65 years | 18
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: age, years] — age in years
  age, years | 35 [26 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Bone Tunnel Diameter
Description: Bone tunnel diameter measured on MRI
Time Frame: 2 years
Population: MRI measurement of tunnel dimensions.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- All Patients: Tunnel expansion after ACL-R occurs early and primarily at the tunnel apertures. Expansion may not affect clinical outcome. Younger age, male sex, and delay from injury to ACL-R may be potential risks for enlargement.
Arm/Group | All Patients
Number analyzed (Participants) | 18
mm | 14.4 (3.8)

2. Other Pre Specified Outcome: Bone Tunnel Cross Sectional Area
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No